CLINICAL TRIAL: NCT04777630
Title: The Neurochemistry and Connectivity in the Brain in Charles Bonnet Syndrome
Brief Title: Neuroscience of Charles Bonnet Syndrome
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID15262; IRAS No: 290078 (Other: Health Regulatory Authority)
Record Dates: First submitted 2021-02-17; First posted 2021-03-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Charles Bonnet Syndrome
Keywords: charles bonnet; visual brain; hallucinations; low vision
MeSH Terms: conditions — Charles Bonnet Syndrome; Hallucinations; Vision, Low | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low vision who experience Charles Bonnet hallucinations: No intervention, observation of neuroimaging and questionnaires
  Interventions: Diagnostic Test: None, neuroimaging
- Patients with low vision who do not experience Charles Bonnet hallucinations: No intervention, observation of neuroimaging and questionnaires
  Interventions: Diagnostic Test: None, neuroimaging

INTERVENTIONS:
Diagnostic Test: None, neuroimaging — Observation only to observe differences in neuroimaging

SUMMARY:
Charles Bonnet Syndrome (CBS) is a condition in which people experience complex visual hallucinations, such as 'Acrobats balancing on bicycles' or 'Spiders crossing meals'. The condition usually occurs in people who have significant vision loss due to eye disease. The aim of this project is to help understand how these hallucinations come about.

In the healthy visual system, the eye provides input to a large area of the brain that performs the computations required to allow us to see the world. There are specialised brain regions responsible for processing of faces, objects, motion and colour. When the eye is no longer working, these parts of the brain lose their input and this may lead to abnormal activity.

Not all people with eye disease and vision loss develop CBS, so the investigators will use magnetic resonance imaging (MRI) to compare the brains of people with and without the condition. In particular the investigators are interested in measuring the levels of chemicals in the visual areas of the brain to see whether they are disrupted in CBS, leading to the hallucinations. It is possible to measure how the different areas of the visual brain are connected together and see whether this is altered in CBS, perhaps with increases in the strength of connection between specialised areas. These measures will be related to questionnaires about hallucinations and vision. This will be done by comparing low vision who experience Charles Bonnet visual hallucinations compared to low vision patients who do not have hallucinations. Assessments will take place at the Wellcome Centre for Integrative Imaging (WIN) based at the John Radcliffe Hospital.

The study will provide insight into the role of the brain in generating CBS hallucinations, helping us to design a larger study and eventually to test whether there are interventions to help improve the condition.

DETAILED DESCRIPTION:
Charles Bonnet Syndrome (CBS) has been reported in people with visual impairment, and is surprisingly common with an estimated prevalence of 10-34% of low vision patients from local audits. It consists of complex visual hallucinations such as seeing snakes rising from people's heads or elephants inside a room (see review, Carpenter, Jolly et al. 2019). Patients experience CBS hallucinations over many years, and although they retain knowledge it is not real, the hallucinations can be frightening and cause considerable distress. Patients with CBS have a lower quality of life compared to patients with vision loss without CBS. Moreover, CBS is under reported due to the fear of being labelled with mental health disease, adding to the negative consequences.

There is currently no established treatment for CBS, with the mainstay of management in low vision clinics revolving around reassurance. Many patients receive inappropriate care from other healthcare practitioners as reported by Judith Potts, founder of Esme's Umbrella, a patient support charity dedicated to Charles Bonnet Syndrome. A clearer understanding of the mechanisms underlying CBS would help to ensure the medical community takes the condition seriously and therefore adequately counsel presenting patients. In addition, understanding the neural mechanisms of CBS can provide a model for investigating how the brain reorganizes in response to sensory impairment and may eventually lead to improvement in the management and treatment of the neurological consequences of eye disease.

Visual processing becomes more complex throughout the pathway from the retina, primary visual cortex to the more specialised processing in higher visual areas. Thus, the complex nature of the hallucinations in CBS (faces, objects, animals), in spite of blurred vision, appears to implicate the higher visual areas in the visual ventral stream that are known to be process objects.

Neurotransmitters are the chemicals that allow communication across the brain. Some neurotransmitters increase the activity in the brain (excitatory) and others reduce activity (inhibitory). A candidate mechanism for CBS from computational modelling is the imbalance of excitation:inhibition: loss of feedforward visual input may give greater prominence to feedback in higher visual areas, causing hallucinations. A recent EEG study has provided experimental support, showing that hyperexcitability of the visual cortex was a key difference between people who have hallucinations versus those who do not. A critical proof of this theory would require measurement of excitatory and inhibitory neurochemicals, glutamate and GABA respectively, in visual areas. This is still outstanding and will be tackled by this study. MRS-imaging is a cutting-edge method to quantify the concentration of neurochemicals in the brain. Rather than providing a single measurement from a large volume of tissue (30x30x30mm), this technique provides high spatial resolution (5x5x20mm) measurements that permits comparison across the visual cortex. MRSI is the only technique that can non-invasively quantify neurochemicals in the living human brain, and MRS-imaging can provide concentrations of the neurotransmitters in multiple locations, which can then be compared across groups.

In summary, based on previous work and the nature of the hallucinations, the investigators predict that patients with CBS likely show 1) changes in the neurotransmitter balance across the visual cortex; 2) increased influence of feedback mechanisms from higher visual areas and 3) abnormal activity in the ventral visual stream to visual stimulation. Our goal is to characterise the visual cortex of CBS patients by using rigorous non-invasive multi-modal MR imaging techniques. Using state-of-the-art methods, the team will measure concentrations of excitatory and inhibitory neurotransmitters, identify changes in connectivity, and measure evoked visual activity in patients with CBS and visually impaired participants without CBS. In addition, the team will obtain clinical evaluation and qualitative assessments of hallucinations.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing & able to give informed consent for participation in the study.
* Male or female, aged 18 - 70 years.
* Reduced vision.

Exclusion Criteria:

* Pre-existing amblyopia or squint.
* Insufficient understanding of written and verbal English to complete safety screening questionnaires.
* Pregnancy or trying to conceive.
* Other neurological problems which may confound the results, e.g. diagnosis of Parkinsons.
* Contraindication to MRI e.g. claustrophobia, presence of metallic implants, a pacemaker, recent surgery etc.
* MR Spectroscopy contraindications e.g. use of antidepressants or antipsychotic medication, frequent cigarette and alcohol consumption. This is defined as no more than one cigarette per day within the past 3 months, and no alcohol use within 3 days prior to scanning.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be two cohorts of participants. Cohort one will consist of low vision (as defined clinically) patients who experience visual hallucinations and cohort two will consist of low vision patients who do not experience visual hallucinations. Male and female adults will be included.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
To assess changes in neurotransmitter balance across the visual cortex in patients with hallucinations compared to without hallucinations using MRSI. | 1 day
  Comparison of neurotransmitter concentrations in different areas of the visual cortex. Correlation of these with the results of the questionnaires about hallucinations.

SECONDARY OUTCOMES:
To characterise the connectivity of visual areas across the brain in patients with hallucinations compared to without hallucinations (resting state and diffusion MRI). | 1 day
  Connectivity between visual centres (resting state MRI) and microstructural properties of the white matter from diffusion MRI (FA and MD).
To assess functional changes in the ventral visual stream in patients with hallucinations compared to without hallucinations (functional MRI). | 1 day
  Difference in Blood oxygenation level dependent (BOLD) response to simple and complex stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Jasleen K Jolly, DPhil, Principal Investigator — University of Oxford; Betina Ip, DPhil, Study Chair — University of Oxford; Holly Bridge, DPhil, Study Director — University of Oxford
Locations (2):
- United Kingdom (2):
  - Vision and Eye Research Institute, Cambridge
  - Wellcome Centre for Integrative Neuroimaging, Oxford

IPD SHARING:
Plan to Share IPD: Undecided